CLINICAL TRIAL: NCT01577693
Title: An Open-label, Single Dose, Randomized, Two-period Crossover Study to Investigate the Bioavailability of a Novel Dosage Form of Dutasteride in Healthy Male Subjects
Brief Title: Study to Compare the Bioavailability of Dutasteride Novel Formulation Form to the Soft Gel Capsule Form in Healthy Male Subjects
Acronym: ARI115148
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115148
Record Dates: First submitted 2011-08-11; First posted 2012-04-16 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Prostatic Hyperplasia
Keywords: dutasteride; cross over study; bioavailability
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5 mg novel dose form (test) (Experimental): 0.5 mg novel dose form (test)
  Interventions: Drug: dutasteride
- 0.5 mg Soft Gel Capsule (Other): 0.5 mg Soft Gel Capsule (reference)
  Interventions: Drug: dutasteride

INTERVENTIONS:
Drug: dutasteride — novel dutasteride
  Arms: 0.5 mg novel dose form (test)
Drug: dutasteride — dutasteride soft gel capsule
  Arms: 0.5 mg Soft Gel Capsule

SUMMARY:
The purpose of this study is to determine the bioavailability of 0.5mg dutasteride novel formulation compared to the currently marketed 0.5mg dutasteride soft gel capsule in fasted healthy male subjects.

DETAILED DESCRIPTION:
The purpose of this study is to determine the bioavailability of 0.5mg dutasteride in a novel formulation compared to the currently marketed 0.5mg dutasteride soft gel capsule in fasted healthy male subjects. This will be an open-label, single dose, randomized, two-period crossover study in healthy male subjects. Subjects will receive a single oral dose 0.5mg novel dutasteride formulation and a single oral dose 0.5mg dutasteride soft gel capsule in a fasted state. Each dose of the study medication will be separated by a 28-day washout period. Blood samples for pharmacokinetic analysis will be taken at regular intervals after dosing. Safety will be assessed by measurement of blood pressure, heart rate, laboratory data, and review of adverse events. The study will enrol approximately 35 healthy male subjects to ensure that 30 subjects complete the study. The study will be conducted in the USA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician.
* Males between 20 and 45 years of age inclusive, at the time of signing the informed consent form.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception.
* Body mass index within the range 18-30 kg/m2 (inclusive); weight range 55-95 kg (inclusive).
* Capable of giving written informed consent.
* Single QTcB < 450 msec.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* History of postural hypotension, dizziness, poor hydration, vertigo, vaso-vagal reactions or any other signs and symptoms of orthostasis.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for human immunodeficiency virus (HIV) antibody.
* Subject is mentally or legally incapacitated.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements.
* History of sensitivity to dutasteride, components thereof or drugs of this class or a history of drug or other allergy.
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* The subject has participated in a clinical trial for 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* A positive pre-study drug/alcohol screen.
* History of regular alcohol consumption.
* Consumption of red wine, grapefruit juice, grapefruit and related hybrids, and jufen grapes.
* The subject has donated blood or blood products in excess of 500 mL within a 56 day period.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-05-12 (Actual); Primary Completion 2011-08-31 (Actual); Study Completion 2011-08-31 (Actual)

PRIMARY OUTCOMES:
Bioavailability | Change from Day 1 (session 1) compared to Day 29 (session 2), predose, .25, .5, .75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72
  To assess the dutasteride relative bioavailability of the of 0.5 mg novel formulation compared with the currently marketed 0.5 mg soft gelatin capsule.

SECONDARY OUTCOMES:
Safety | Changes from screening to 3 months
  Changes in blood pressure and pulse rates, review of number of subjects with adverse events, and changes in clinical laboratory data.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115148 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115148?search=study&search_terms=115148#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 115148 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115148 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115148 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115148 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115148 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115148 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115148 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register